CLINICAL TRIAL: NCT05779579
Title: A Randomized, Double-blind, Placebo-controlled Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics Characteristics and Primary Efficacy of HS-10517 in Chinese Adult Participants
Brief Title: Study of HS-10517 in Chinese Adult Participants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HS-10517-101
Record Dates: First submitted 2023-01-16; First posted 2023-03-22 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: HS-10517; 3CL protease inhibitor; single ascending dose; multiple ascending dose; phase 2 study; dose exploration; Chinese; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HS-10517 Dose 1 (Experimental): Dose level 1 of HS-10517 Tablets，Dose 1
  Interventions: Drug: HS-10517 Dose 1
- HS-10517 Dose 2 (Experimental): Dose level 1 of HS-10517 Tablets，Dose 2
  Interventions: Drug: HS-10517 Dose 2
- HS-10517 Dose 3 (Experimental): Dose level 1 of HS-10517 Tablets，Dose 3
  Interventions: Drug: HS-10517 Dose 3
- HS-10517 Dose 4 (Experimental): Dose level 1 of HS-10517 Tablets，Dose 4
  Interventions: Drug: HS-10517 Dose 4
- Placebo Comparator (Experimental): Dose level A of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10517 Dose 1 — HS-10517 Dose 1+Ritonavir
  Arms: HS-10517 Dose 1
Drug: HS-10517 Dose 2 — HS-10517 Dose 2+Ritonavir
  Arms: HS-10517 Dose 2
Drug: HS-10517 Dose 3 — HS-10517 Dose 3+Ritonavir
  Arms: HS-10517 Dose 3
Drug: HS-10517 Dose 4 — HS-10517 Dose 4+Ritonavir
  Arms: HS-10517 Dose 4
Drug: Placebo — Dose level A of placebo
  Arms: Placebo Comparator

SUMMARY:
A Phase I/II, randomized, double-blind, placebo-controlled study to evaluate safety, tolerability, pharmacokinetics and primary efficacy of HS-10517 in Chinese adult participants.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for SAD, MAD and SE：

* Subjects should fully understand the content, process and possible adverse reactions of the study, and voluntarily sign the informed consent form;
* The age at the time of signing the informed consent is between 18 and 45 years old (including the critical value)
* Subjects with negative COVID-19 nucleic acid detection in screening period;
* The body mass index (BMI=body weight [kg]/height2 [m2]) at screening is 19~27kg/m2 (including the critical value), and the weight of men is ≥ 50kg, and that of women is ≥ 40kg;
* The blood pregnancy test of female subjects in the screening period and the baseline period is negative;
* Female subjects must agree to take effective contraceptive measures from the date of signing the informed consent form to 30 days after the last administration:

  1. Those with fertility: from the date of signing the informed consent form to 30 days after the last administration, ① avoid pregnancy, ② if having sex with the opposite sex, agree to continue to use one or more forms of effective contraception (such as verified intrauterine devices, bilateral tubal ligation or correct use of condoms, excluding any form of hormonal contraceptives). If the male partner has undergone an effective sterilization operation, additional effective contraception measures should be taken when the sperm is uncertain);
  2. Non-fertility: ① Postmenopausal (spontaneous amenorrhea ≥ 12 months, or spontaneous amenorrhea ≥ 6 months and FSH>40 IU/L, without other obvious pathological or physiological reasons) before screening; Or ② documented surgical sterilization (such as hysterectomy, bilateral salpingectomy or bilateral oophorectomy, etc.);
* Male subjects (including their female partners) must agree to take effective contraceptive measures from the date of signing the informed consent form to 30 days after the last administration:

  1. Those who are fertile must agree to use condoms correctly. If their female partners are women of child-bearing age and have fertility (have not undergone hysterectomy, bilateral salpingectomy or bilateral oophorectomy and have no medical proven ovarian failure), their female partners must take effective contraceptive measures (such as oral/injection/vaginal or implantable hormone contraceptives, or other physical barrier, surgery and other female contraceptive methods) within 30 days after the last administration;
  2. Those who are infertile, such as those who have undergone effective sterilization operations, take additional effective contraceptive measures when they are not sure whether they have sperm);
* Male subjects agree to avoid donating sperm within 30 days from the initiation of drug administration until the last administration.

Inclusion Criteria for Phase II dose exploration:

* Subjects should fully understand the content, process and possible adverse reactions of the study, and voluntarily sign the informed consent form;
* The age at the time of signing the informed consent is ≥ 18 years old;
* In the first 2 days (48 hours) before randomization, COVID-19 nucleic acid detected by RT-PCR is positive;
* During the screening period, the subject is assessed by the research doctor as a patient with mild to moderate COVID-19 infection;
* During the screening period, the subject is assessed by the research doctor and show symptoms/signs of COVID-19 infection for the first time within 2 days before randomization;
* At least one of targeted COVID-19 symptoms exists within the first 24 hours of randomization and meets the corresponding severity;
* Female subjects must agree to take the drug from the date of signing the informed consent form to 30 days after the last administration; Effective contraceptive measures:

Those with fertility: from the date of signing the informed consent form to 30 days after the last administration, ① avoid pregnancy, ② if having sex with the opposite sex, agree to continue to use one or more forms of effective contraception (such as verified intrauterine devices, bilateral tubal ligation or correct use of condoms, excluding any form of hormonal contraceptives). If the male partner has undergone an effective sterilization operation, additional effective contraception measures should be taken when the sperm is uncertain);

* Male subjects (including their female partners) agree to take effective contraceptive measures from the date of signing the informed consent form to 30 days after the last administration:

  1. Those who are fertile must agree to use condoms correctly. If their female partners are women of child-bearing age and have fertility (have not undergone hysterectomy, bilateral salpingectomy or bilateral oophorectomy and have no medical proven ovarian failure), their female partners must take effective contraceptive measures (such as oral/injection/vaginal or implantable hormone contraceptives, or other physical barrier, surgery and other female contraceptive methods) within 30 days after the last administration
  2. Those who are infertile, such as those who have undergone effective sterilization, take additional effective contraceptive measures when they are not sure whether they have sperm).
* The pregnancy test of female subjects in the screening period and the baseline period is negative;
* Male subjects agree to avoid donating sperm within 30 days from the start of administration until the last administration

Exclusion Criteria of SAD, MAD and SE:

* According to the judgment of the principal investigator, the participant is accompanied with suspected COVID-19 related clinical symptoms/signs;
* During screening, those who are judged to be clinically significant by the principal investigator through medical history inquiry, physical examination, vital signs, blood oxygen saturation (SpO2), laboratory examination, 12-lead electrocardiogram (ECG), abdominal ultrasound, chest X-ray examination, etc;
* Participants with clinically significant diseases (such as neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal muscle system, endocrine and metabolic system, blood system, skin disease, immune system, tumor, etc.) are evaluated by the researcher as not suitable for this study;
* Previous major surgery, or according to the judgment of the principal investigator, there is any physiological or disease or condition that may affect the absorption of the study drug (such as gastrectomy, cholecystectomy, enterotomy, etc.);
* According to the judgment of the principal investigator, there is any physical or psychological disease or condition that may increase the risk of the test, affect the compliance of the subject with the other case, or affect the subject's completion of the test;
* Within 2 weeks or 5 half-life (whichever is longer) before screening, and during the whole study period, it is expected to take any medicine and health care products, including prescription drugs, over-the-counter drugs and Chinese herbal medicine (including oral contraceptives, external spermicide, drugs with systemic therapeutic effects through percutaneous absorption and St. John's wort);
* Participants have participated in any clinical study or taken study drugs within 3 months before screening;
* Have a history of vaccination within 30 days before screening, or plan to have a vaccination throughout the study period;
* Difficult in blood sample collection, unable to tolerate multiple venous blood collection and any contraindication of blood sample collection;
* Large amount of blood loss or donation (more than 250mL) within 3 months before screening;
* At screening, 12-lead ECG is abnormal and had clinical significance according to the judgment of the researcher, such as the QT interval (QTcB) corrected by Bazett (formula QT/RR0.5), the absolute value of QTcB in males is more than 450ms, and the absolute value of QTcB in females is more than 470ms;
* When screening, endogenous creatinine clearance rate is less than 80mL/min, according to Cockcroft-Gault formula: endogenous creatinine clearance rate (mL/min)=(140 - age) × body weight (kg) 72 × serum creatinine concentration (mg/dL) (female × 0.85);
* During the screening period and/or the baseline period, the blood pressure and pulse are within the following range: systolic blood pressure <90 mmHg or ≥ 140 mmHg, diastolic blood pressure <60 mmHg or ≥ 90 mmHg, pulse <55 bpm or >100 bpm;
* Have a history of drug dependence or drug abuse in the past, or have a positive urine drug test during screening;
* Those who have a history of severe allergy to drugs, food and articles (including allergy to latex, dust mites, pollen, etc.), or are known to be allergic to the test drug ingredients;
* Within 2 weeks before screening, dieting or receiving dietary treatment for whatever reason, or major changes in dietary habits;
* Have a history of alcoholism in the past (drinking more than 14 units of alcohol per week on average), or drink more than 14 units of alcohol per time in the past two weeks (1 unit=285mL of beer, 25mL of spirits, 125mL of wine), or cannot stop drinking alcohol products during the test; Or positive alcohol breath test during screening;
* Those who smoke more than 5 cigarettes per day on average in the three months before screening, or who cannot stop using any tobacco products during the test;
* Within 2 weeks before screening, subjects ingested foods that may affect drug metabolism, such as grapefruit juice;
* The average daily intake of coffee, tea, cola or other caffeinated drinks exceeds 6 cups (about 250mL per cup) within 3 months before screening;
* Those who have difficulty swallowing solid preparations such as tablets;
* Female subjects are in pregnancy or lactation at the time of screening;
* This study may not be completed due to other reasons or the researcher judges that it is not suitable for participants.

Exclusion Criteria for Phase II dose exploration:

* The medical condition indicates that COVID-19 causes clinical signs of severe systemic diseases, such as respiratory rate ≥ 30 times/minute, heart rate ≥ 125 times/minute, blood oxygen saturation (SpO2) ≤ 93% or PaO2/FiO2<300 mmHg within 24 hours before randomization (under indoor air conditions at rest), and it is urgent or expected to require nasal high-flow oxygen therapy or non-invasive positive pressure ventilation, invasive mechanical ventilation or ECMO.
* According to the judgment of the researcher, the medical condition suggests that COVID-19 may develop into severe/critical status in the next 48 hours;
* Other than COVID-19, suspected or confirmed acute systemic infection (such as combined influenza and bacterial infection) may interfere with the evaluation of the research intervention response.
* Known history of active liver disease (excluding nonalcoholic fatty liver), including acute or chronic active hepatitis B or C, primary biliary cirrhosis, Child-Pugh grade B or C or acute liver failure.
* The patient is undergoing dialysis or is known to have moderate to severe renal damage (that is, within 6 months before the screening visit, the CKD-EPI formula based on serum creatinine eGFR < 45mL/min/1.73m2).
* They received anti-COVID-19 drugs (excluding NSAIDs) within 14 days before randomization.
* Has received (within 30 days before randomization or within the half-life of 5 drugs, whichever is longer) or is expected to receive COVID-19 monoclonal antibody or COVID-19 convalescence plasma treatment during the study period.
* Any anti-COVID-19 vaccine was inoculated within 3 months before randomization.
* Subjects who have to use potent CYP3A4/5 inhibitors and/or potent CYP3A4/5 inducers from 7 days before screening to 7 days after the last administration for various reasons.
* Subjects have major diseases (such as acute myocardial infarction, stroke, malignant tumor, etc.) within 30 days before signing the informed consent form;
* Those who have difficulty swallowing solid preparations such as tablets;
* At the time of screening, the female subjects are in pregnancy or lactation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AE), serious adverse events (SAE) and adverse events leading to withdrawal from the trial and the correlation with the investigational drug in single ascending dose (SAD) | Day 1 to Day 5
  The definition of adverse event [AE] is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The definition of serious adverse event [SAE] is any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.
Number of participants with clinically significant change from baseline in vital signs in SAD | Day 1 to Day 5
Number of participants with clinically significant change from baseline in 12-lead electrocardiogram (ECG) findings in SAD | Day 1 to Day 5
  Criteria for clinically significant changes in 12-lead ECG are defined as: a postdose QTc interval increase by ≥30 msec from the baseline and is >450 msec; or an absolute QTc value is ≥500 msec for any scheduled 12-lead ECG.
Number of participants with clinically significant abnormalities in laboratory examination in SAD | Day 1 to Day 5
Number of participants with clinically significant abnormalities in physical examination in SAD | Day 1 to Day 5
The incidence and severity of adverse events (AE), serious adverse events (SAE) and adverse events leading to withdrawal from the trial and the correlation with the investigational drug in multiple ascending dose (MAD) | Day 1 to Day 14
  The definition of adverse event [AE] is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The definition of serious adverse event [SAE] is any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.
Number of participants with clinically significant change from baseline in vital signs in MAD | Day 1 to Day 14
Number of participants with clinically significant change from baseline in 12-lead electrocardiogram (ECG) findings in MAD | Day 1 to Day 14
  Criteria for clinically significant changes in 12-lead ECG are defined as: a postdose QTc interval increase by ≥30 msec from the baseline and is >450 msec; or an absolute QTc value is ≥500 msec for any scheduled 12-lead ECG.
Number of participants with clinically significant abnormalities in laboratory examination in MAD | Day 1 to Day 14
Number of participants with clinically significant abnormalities in physical examination in MAD | Day 1 to Day 14
The incidence and severity of adverse events (AE), serious adverse events (SAE) and adverse events leading to withdrawal from the trial and the correlation with the investigational drug in supratherapeutic exposure (SE) | Day 1 to Day 13
  The definition of adverse event [AE] is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The definition of serious adverse event [SAE] is any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.
Number of participants with clinically significant change from baseline in vital signs in SE | Day 1 to Day 13
Number of participants with clinically significant change from baseline in 12-lead electrocardiogram (ECG) findings in SE | Day 1 to Day 13
  Criteria for clinically significant changes in 12-lead ECG are defined as: a postdose QTc interval increase by ≥30 msec from the baseline and is >450 msec; or an absolute QTc value is ≥500 msec for any scheduled 12-lead ECG.
Number of participants with clinically significant abnormalities in laboratory examination in SE | Day 1 to Day 13
Number of participants with clinically significant abnormalities in physical examination in SE | Day 1 to Day 13
Percentage of participants with a negative RT-PCR test through day 5-modified intent-to-treat (mITT) population. | Day 1 to Day 5

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) in SAD | Day 1 to Day 5
  The maximum observed plasma concentration [Cmax] is estimated based on the plasma concentrations.
Time for Cmax (tmax) in SAD | Day 1 to Day 5
  Tmax was summarized by dosing regimen. It was observed directly from data as time of first occurrence.
Area under the concentration time profile from time 0 to the time of last quantifiable plasma concentration (AUC0-last) in SAD | Day 1 to Day 5
  AUC0-last is summarized by dosing regimen and determined by linear/log trapezoidal method.
Area under the concentration time profile from time 0 to infinity (AUC0-inf) in SAD | Day 1 to Day 5
  AUC0-inf is summarized by dosing regimen and determined by linear/log trapezoidal method.
Terminal rate constant (λz) in SAD | Day 1 to Day 5
Terminal half-life (t1/2) in SAD | Day 1 to Day 5
Apparent clearance (CL/F) in SAD | Day 1 to Day 5
Apparent volume of distribution (Vd/F) in SAD | Day 1 to Day 5
Mean residence time (MRT) in SAD symptoms to the sustained clinical resolution within 28 days（Phase II） | Day 1 to Day 5
Maximum plasma concentration (Cmax) in first dose of MAD | Day 1 to Day 14
  The maximum observed plasma concentration [Cmax] is estimated based on the plasma concentrations.
Time for Cmax (tmax) in first dose of MAD | Day 1 to Day 14
  Tmax was summarized by dosing regimen. It was observed directly from data as time of first occurrence.
Area under the concentration time profile from time 0 to 24 hours in first dose of MAD | Day 1 to Day 14
  AUC0-24 is summarized by dosing regimen and determined by linear/log trapezoidal method.
Area under the concentration time profile from time 0 to 12 hours in first dose of MAD | Day 1 to Day 14
  AUC0-12 is summarized by dosing regimen and determined by linear/log trapezoidal method.
Maximum plasma concentration at steady state (Css,max) in last dose of MAD | Day 1 to Day 14
Time for Cmax at steady state (tss,max) in last dose of MAD | Day 1 to Day 14
Minimum plasma concentration at steady state (Css,min) in last dose of MAD | Day 1 to Day 14
Area under the concentration time profile in one dosing interval at steady state (AUCss) in last dose of MAD | Day 1 to Day 14
Apparent clearance at steady state (CLss/F) in last dose of MAD | Day 1 to Day 14
Degree of accumulation after multiple doses (RAC, including RAUC and RCmax) in last dose of MAD | Day 1 to Day 14
Maximum plasma concentration (Cmax) in SE | Day 1 to Day 13
  The maximum observed plasma concentration [Cmax] is estimated based on the plasma concentrations.
Time for Cmax (tmax) in SE | Day 1 to Day 13
  Tmax was summarized by dosing regimen. It was observed directly from data as time of first occurrence
Area under the concentration time profile from time 0 to the time of last quantifiable plasma concentration (AUC0-last) in SE | Day 1 to Day 13
  AUC0-last is summarized by dosing regimen and determined by linear/log trapezoidal method
Area under the concentration time profile from time 0 to infinity (AUC0-inf) in SE | Day 1 to Day 13
  AUC0-inf is summarized by dosing regimen and determined by linear/log trapezoidal method
Terminal rate constant (λz) in SE | Day 1 to Day 13
Terminal half-life (t1/2) in SE | Day 1 to Day 13
Apparent clearance (CL/F) in SE | Day 1 to Day 13
Apparent volume of distribution (Vd/F) in SE | Day 1 to Day 13
Mean residence time (MRT) in SE | Day 1 to Day 13
Time to sustained resolution of 11 COVID-19 symptoms within 28 days | Day 1 to Day 28
  All of the 11 COVID-19-related symptoms consist of stuffy or running nose, sore throat, shortness of breath, cough, muscle or body aches, headache, chills or shivering, feeling hot or feverish, nausea, vomiting, diarrhea. Sustained resolution is defined as when all targeted symptoms were scored as 0 for 2 consecutive days.
Change of viral load over time compared to baseline | Day 1 to Day 28
Time to the first negative RT-PCR test | Day 1 to Day 28
Virological response at each time point after randomization | Day 1 to Day 28
  virological response means the rate of negative RT-PCR test
Time to sustained alleviation of 11 targeted COVID-19 signs/symptoms within 28 days | Day 1 to Day 28
  Sustained alleviation of 11 targeted COVID-19 signs/symptoms was defined as the event occurring on the first 2 consecutive days when 11 targeted symptoms scored as moderate or severe at the time of enrollment were scored as mild or absent and those scored mild or absent at the time of enrollment were scored as absent. The first day of the 2 consecutive-day period was considered date of first event. Time to sustained recovery [event] was calculated as first event date minus first dose date plus 1, for participants with event. For participants who completed Day 28 or discontinued the study before Day 28 without sustained resolution [censored], time was calculated as censoring date [last date on which symptom recovery was assessed] minus first dose date plus 1 or Day 25 whichever occurred first.
Time to sustained resolution of each targeted COVID-19 symptom | Day 1 to Day 28
Change of the score of each COVID-19 symptom | Day 1 to Day 28
  11 targeted COVID-19 related clinical symptoms) from baseline up to 28 days
Proportion of severe cases within 28 days | Day 1 to Day 28
  All 4 inclusion criteria should be met in severe cases: positive RT-PCR test; respiratory distress [respiratory rate > 30 times/min]; hypoxia [resting oxygen saturation < 93% or arterial partial pressure of oxygen / oxygen concentration < 300 mmHg]; COVID-19 featured lung lesions in chest X-ray image.
The plasma concentration of HS-10517 in COVID-19 patients in phase II study | Day 1 to Day 7
Population apparent clearance (CL/F) of COVID-19 patients in phase II study | Day 1 to Day 7
Population apparent volume of distribution (Vd/F) of COVID-19 patients in phase II study | Day 1 to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No